CLINICAL TRIAL: NCT03767946
Title: MTBVAC in Newborns: Epidemiological Study In Tuberculosis-Endemic Regions of Sub-Saharan Africa
Brief Title: Epidemiological Study In Tuberculosis-Endemic Urban Area in Senegal
Acronym: MTBVAC-EPI
Status: Completed | Type: Observational
Sponsor: Biomedical Research Center EPLS (Other)
Collaborators: Biofabri, S.L (Industry); TuBerculosis Vaccine Initiative (Other); Universidad de Zaragoza (Other); University of Cape Town (Other); Institut Pasteur de Madagascar (Other)
Responsible Party: Principal Investigator, Gilles Riveau, PharmD, PhD, CEO, Biomedical Research Center EPLS
Other Study IDs: RIA2016V-1637
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Quantiferon Gold Plus test; Tuberculosis in children; SENEGAL; MTBVAC
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for Quantiferon Gold Plus assay
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Children both genders according to age:
  *1-year old children (12 months -1/+4 months); n=125 at the date of recruitment.
  Interventions: Diagnostic Test: Quantiferon Gold Plus Test
- Group 2: Children both genders according to age:
  *2-year-old children (24 months -1/+4 months); n=125 at the date of recruitment.
  Interventions: Diagnostic Test: Quantiferon Gold Plus Test
- Group 3: Children both genders according to age:
  *5-year old children (60 months +/- 6 months); n=125 at the date of recruitment.
  Interventions: Diagnostic Test: Quantiferon Gold Plus Test
- Group 4: Children both genders according to age:
  *12-years old children (12 years old +/- 6 months); n=125 at the date of recruitment.
  Interventions: Diagnostic Test: Quantiferon Gold Plus Test

INTERVENTIONS:
Diagnostic Test: Quantiferon Gold Plus Test — Small volume of whole blood incubated with specific TB antigen and then dosage of Interferon gamma production.

SUMMARY:
A cross-sectional childhood M. tuberculosis infection survey of age-specific rates (defined by positivity to the test QuantiFERON-TB Gold Plus) will be conducted in Senegal to collect information on the local TB endemic to inform site selection, sample size, and recruitment strategies for a future efficacy trial of vaccine candidate MTBVAC in young children.

DETAILED DESCRIPTION:
MTBVAC is a new TB vaccine candidate based on an attenuated clinical isolate of M. tuberculosis. The clinical development consortium of this EDCTP program is preparing for future years an MTBVAC efficacy trial by setting up a network of three African sites in South Africa, Senegal and Madagascar. Each site has established an operational clinical research infrastructure. As a first step, Senegal site needs to collect crucial epidemiological data on TB in children, to allow a rapid transition to a phase 3 trial in infants.

The primary objective is to estimate the prevalence of TB infection by the QuantiFERON-TB Gold Plus technique in 500 children splined in 1-year, 2-year, 5-year, and 12-year-old age groups living in the study area (Saint Louis, Senegal).

Secondary objectives are:

* To study the socio-demographic characteristics, the vaccination history of each subject and the possible tuberculous contacts he has.
* To map selected populations (from GPS residence data) according to the status (infected or uninfected) of each subject.
* To ensure the orientation of children found positive by the QuantiFERON-TB Gold Plus test for care and follow-up related to the TB diagnosis and treatment at one of the Health Centers (THC) located in the study areas.
* To estimate the number of tuberculosis cases detected in children aged up to 12 years and resident in the study area from THC registries and data from the National Tuberculosis Control Plan (PNB).

ELIGIBILITY:
Inclusion Criteria:

* Children resident in the study area (St Louis City)
* Obtaining written consent from one of the parents / guardians.
* Children meeting one the following age criterion:

  * 1-year old child (12 months -1/+4 months);
  * 2-year-old child (24 months -1/+4 months);
  * 5-year old child (60 months +/-6 months);
  * 12-year old child (12 years old +/-6 months);

Exclusion Criteria:

* Child resident outside the study area.
* Participation refusal by one of the parents / guardians.
* Objection of the child belonging to the 12-year old group.
* Child with a known chronic pathology (severe asthma, epilepsy, type 1 diabetes, severe immunosuppression ...)
* Child considered by the Principal Investigator as medically unfit to participate in the study.

Ages: 11 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A convenience sample taking into account the constraints related to the QuantiFERON-TB Gold Plus technique was chosen. One hundred and twenty-five (125) children per age group (1 year, 2 years, 5 years and 12 years) will be included. In total, 500 children will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Tuberculosis prevalence in children living in urban area in Senegal. | 2 days
  To estimate the prevalence of TB infection by QuantiFERON-TB Gold Plus test in children aged 1 year, 2 years, 5 years and 12 years in the city of Saint Louis, Senegal. Blood samples are incubated with TB antigens and then Interferon Gamma production is evaluated by Elisa.

SECONDARY OUTCOMES:
health survey of the cohort | 2 hours
  To carry out a standard questionnaire of the mother of the child included about his vaccinations, the conditions of the child's life and the tuberculous history of his relatives.

CONTACTS AND LOCATIONS:
Overall Officials: Amadou T LY, Principal Investigator — Biomedical Research Center EPLS
Locations (1):
- Biomedical Research Center EPLS, Saint-Louis, France

IPD SHARING:
Plan to Share IPD: Undecided
A plan to make individual participant data (IPD) collected in this study, including data dictionaries, available to other researchers will be defined in the next semester by partners of the project.

REFERENCES:
- [Background] Arbues A, Aguilo JI, Gonzalo-Asensio J, Marinova D, Uranga S, Puentes E, Fernandez C, Parra A, Cardona PJ, Vilaplana C, Ausina V, Williams A, Clark S, Malaga W, Guilhot C, Gicquel B, Martin C. Construction, characterization and preclinical evaluation of MTBVAC, the first live-attenuated M. tuberculosis-based vaccine to enter clinical trials. Vaccine. 2013 Oct 1;31(42):4867-73. doi: 10.1016/j.vaccine.2013.07.051. Epub 2013 Aug 17. PMID 23965219
- [Background] Marinova D, Gonzalo-Asensio J, Aguilo N, Martin C. MTBVAC from discovery to clinical trials in tuberculosis-endemic countries. Expert Rev Vaccines. 2017 Jun;16(6):565-576. doi: 10.1080/14760584.2017.1324303. Epub 2017 May 12. PMID 28447476
- [Background] Cuevas LE, Browning R, Bossuyt P, Casenghi M, Cotton MF, Cruz AT, Dodd LE, Drobniewski F, Gale M, Graham SM, Grzemska M, Heinrich N, Hesseling AC, Huebner R, Jean-Philippe P, Kabra SK, Kampmann B, Lewinsohn D, Li M, Lienhardt C, Mandalakas AM, Marais BJ, Menzies HJ, Montepiedra G, Mwansambo C, Oberhelman R, Palumbo P, Russek-Cohen E, Shapiro DE, Smith B, Soto-Castellares G, Starke JR, Swaminathan S, Wingfield C, Worrell C. Evaluation of tuberculosis diagnostics in children: 2. Methodological issues for conducting and reporting research evaluations of tuberculosis diagnostics for intrathoracic tuberculosis in children. Consensus from an expert panel. J Infect Dis. 2012 May 15;205 Suppl 2(Suppl 2):S209-15. doi: 10.1093/infdis/jir879. Epub 2012 Apr 3. PMID 22476719
- [Result] Nemes E, Rozot V, Geldenhuys H, Bilek N, Mabwe S, Abrahams D, Makhethe L, Erasmus M, Keyser A, Toefy A, Cloete Y, Ratangee F, Blauenfeldt T, Ruhwald M, Walzl G, Smith B, Loxton AG, Hanekom WA, Andrews JR, Lempicki MD, Ellis R, Ginsberg AM, Hatherill M, Scriba TJ; C-040-404 Study Team and the Adolescent Cohort Study Team. Optimization and Interpretation of Serial QuantiFERON Testing to Measure Acquisition of Mycobacterium tuberculosis Infection. Am J Respir Crit Care Med. 2017 Sep 1;196(5):638-648. doi: 10.1164/rccm.201704-0817OC. PMID 28737960